CLINICAL TRIAL: NCT01604759
Title: Evaluation of Polarized Reflectance Spectroscopy for Detection of High-risk Oral Lesions
Brief Title: Polarized Reflectance Spectroscopy for Oral Lesions
Acronym: PolProbe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: M.D. Anderson Cancer Center (Other); University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H10-01313; 5RO1EB00354004 (PC-1) (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2010-11-03; First posted 2012-05-24 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Oral Cancer
Keywords: Mouth Neoplasms; Mouth Diseases
MeSH Terms: conditions — Mouth Neoplasms; Mouth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Polarized probe measurement. (Other): All patients belong under this arm as all will be measured by the polarized probe and the data will be compared to the biopsy site's pathology results.
  Interventions: Device: Polarized Reflectance Spectroscopy System

INTERVENTIONS:
Device: Polarized Reflectance Spectroscopy System — Fiber optic probe designed to measure polarized reflectance spectroscopy will be used to gather data from all study participants.
  Other Names: Polarized Reflectance Spectroscopy System.; Research device developed at MD Anderson Cancer Centre, Dept of Imaging Physics specifically for this study.

SUMMARY:
In this study the investigators are conducting research to determine whether a new optical device using polarization reflectance spectroscopy can help doctors or dentists identify abnormalities in the mouth that require follow-up. To establish this, measurements are needed from a large number of individuals with different abnormalities in their mouth.

The investigators believe the proposed approach has potential to improve and enable mass screening for precancerous and early cancers of the oral cavity by improving the predictive value of oral cavity exams, particularly for less experienced practitioners.

The information from this study will be compared to results from the pathology report of the tissue taken from your mouth.

Hypothesis:

1. Polarized reflectance spectroscopy can distinguish high-risk oral lesion from normal and reactive oral lesions.
2. Polarized reflectance spectroscopy can capture low-grade oral lesions that have characteristics associated with a high risk of progression to cancer.

DETAILED DESCRIPTION:
The clinician will place a fiber-optic probe designed to measure the polarized reflectance spectra over the visible optical region on a site of interest in the subject's mouth, including lesional mucosa, normal adjacent and contralateral mucosa. The site for placement of the probe will be determined by the examiner, an experienced Oral Pathologist. The probe examination will take no more than 15 minutes in addition to the subject's appointment time for their routine visits.

A 4um unstained tissue section from surgery or biopsy, part of their scheduled care, will be requested for quantitative histological analysis. The morphometric parameters obtained from polarized reflectance measurements will be compared with the histology and quantitative pathology (nuclear phenotype score) from the tissue sections from the lesion. The collected spectra data from normal looking areas from adjacent normal looking mucosa and contralateral mucosa will be used to determine patient to patient variation in the polarized reflectance of oral mucosa.

ELIGIBILITY:
Inclusion Criteria:

* You attend the Dental Department at the British Columbia Cancer Agency
* You have an abnormal lesion in the mouth
* You fully understand the study and give your informed consent to participate as demonstrated by signing this consent form

Exclusion Criteria:

* You are under the age of 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To use the spectroscopic data collected to create a model for normal, dysplastic and cancerous tissue. | 2 years
  The goals of the statistical analysis will be to determine an appropriate model for predicting whether the lesion is normal or abnormal (dysplasia or carcinoma) based on spectroscopic characteristics. The investigators will estimate sensitivity and specificity of the predictions made by the model and compare this to sensitivity and specificity of standard white light clinical examination currently used in clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Poh, M.D. Ph.D, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia, Canada